CLINICAL TRIAL: NCT03810144
Title: Impact of Guided Care With the Vectra Multi-biomarker Disease Activity (MBDA) Blood Test on Clinical Outcomes and Pharmaceutical Utilization in Patients With Rheumatoid Arthritis: A Prospective, Randomized Study
Brief Title: Impact of Guided Care With the Vectra Multi-biomarker Disease Activity (MBDA) Blood Test
Acronym: CareFirst
Status: Completed | Type: Observational
Sponsor: Sequenom, Inc. (Industry)
Collaborators: Laboratory Corporation of America (Industry)
Responsible Party: Sponsor
Other Study IDs: 128-CL-01
Record Dates: First submitted 2018-12-26; First posted 2019-01-18 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vectra Guided: For patients in the guided care arm, treating physicians will receive the Vectra MBDA Test score prior to the patient visit and will have a set of guidance for decision-making based on these scores. Treating physicians will be strongly encouraged to follow the guidance but will not be required to do so. For test results to be available at the time of each visit in the MBDA guided treatment arm, blood testing will be performed 7-10 days before the visit.
  Interventions: Genetic: Vectra MBDA Test
- Usual Care: For patients in the UC arm, treating physicians will not have access to MBDA scores until the end of the study.

INTERVENTIONS:
Genetic: Vectra MBDA Test — Vectra Guided versus Usual Care
  Groups: Vectra Guided

SUMMARY:
Nine months multi-center prospective, randomized observational study, two arm trial to evaluate the effect of MBDA score-guided care on disease activity and medical costs.

DETAILED DESCRIPTION:
Nine months multi-center prospective, randomized observational study, two arm trial to evaluate the effect of MBDA score-guided care on disease activity and medical costs. To investigate whether treatment decisions guided by MBDA scores result in reduced disease activity and overall medical cost among patients with RA relative to usual care (UC).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign an informed consent form (ICF)
* Age at least 18 years old at screening visit
* Diagnosed with RA according to 1987 or 2010 criteria of the American College of Rheumatology
* Actively managed by a CareFirst health care practitioner
* Currently taking one or more biologic and/or non-biologic DMARDs listed in Appendix 2
* Currently has CareFirst medical coverage

Exclusion Criteria:

* Active infection
* History of malignancy within the past 5 years or any evidence of persistent malignancy, except fully excised basal cell or squamous cell carcinomas of the skin, or cervical carcinoma in situ that has been treated or excised in a curative procedure
* Current enrollment in another clinical trial
* On non-biologic DMARD monotherapy or combination therapy with stable disease for ≥6 months
* Any condition or circumstance that makes it likely the patient will not be able to complete the 9-month trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with RA who are currently taking one or more non-biologic DMARD and/or biologic DMARD listed in Appendix 2.
Sampling Method: Non-Probability Sample
Enrollment: 444 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-10-16 (Actual)

PRIMARY OUTCOMES:
Mean MBDA Score | Baseline to 9 months
  Change in disease activity from baseline to month 9 as measured by mean MBDA score.
  MBDA Score stands for the Vectra multi-biomarker disease activity (MBDA) blood test.
  Scale: Low (>30); Moderate (30-44); High (>44)

SECONDARY OUTCOMES:
Changes in Overall Medical Costs | Baseline to 1 year
  Changes in overall medical costs, RA-related medical costs, pharmacy costs, RA treatment medication costs, and biologic DMARD medication costs from baseline to one year, as defined in Appendix 2.
Medical Utilization | Baseline to 1 year
  Medical utilization metrics (admissions, readmissions, emergency room visits, physician visits, etc.).
Proportion of Patients who Showed a Response to Medication | Baseline to month 9
  Proportion of patients who showed a response to medication, defined as a decrease in MBDA score of at least 8 from baseline to month 9.
Pharmacy Utilization | Baseline to 1 year
  Pharmacy utilization metrics (days' supply, prescriptions, etc.).
Treatment Adherence | Baseline to 1 year
  Treatment adherence metrics measured according to medical possession ratio and time to discontinuation.

OTHER OUTCOMES:
Proportion of Patients with Non-High MBDA Scores | Baseline to month 9
  Proportion of patients with non-high (≤44) MBDA scores from baseline to month 9.
Overall Medical Costs | Baseline to 1 year
  Overall medical costs, pharmacy costs, RA treatment medication costs, and biologic DMARD medication costs (Appendix 2) from baseline to one year according to:
  1. Baseline MBDA score category (low <30, moderate 30-44, high >44).
  2. Whether treatment decisions were consistent with the MBDA score-based treatment guidance in Appendix 1 (guided treatment arm only).
  3. Whether MBDA score category changed from baseline to month 9.
  4. Whether biologic DMARD use was tapered.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Hitraya, MD, Study Director — Consultant
Locations (11):
- United States (11):
  - Annapolis Rheumatology LLC, Annapolis, Maryland
  - Lifebridge Sinai Hospital of Baltimore, Baltimore, Maryland
  - Rheumatology Associates of Baltimore LLC, Baltimore, Maryland
  - Nasseri Clinic of Arthritis & Rheumatic Diseases, LLC., Catonsville, Maryland
  - Arthritis Care Specialists of Maryland, Columbia, Maryland
  - Klein & Associates, Cumberland, Maryland
  - Mid-Atlantic Rheumatology, Glen Burnie, Maryland
  - Arthritis & Pain Associates of PG County, Greenbelt, Maryland
  - Klein & Associates, Hagerstown, Maryland
  - MedStar Shah Medical Group, Hollywood, Maryland
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland